CLINICAL TRIAL: NCT01006525
Title: Abuse Liability Associated With Chronic Hypnotic Use
Brief Title: Safety and Efficacy of Chronic Hypnotic Use
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Timothy Roehrs, Ph.D., Henry Ford Health System
Other Study IDs: R01DA017355 (NIH)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Insomniacs: Primary insomniacs, ages 21-70, in good general health.
  Interventions: Drug: zolpidem

INTERVENTIONS:
Drug: zolpidem — placebo or zolpidem (10mg)daily for one year
  Other Names: zolpidem (Ambien)

SUMMARY:
The purpose of the study is to determine how safe and effective it is for people with insomnia to use zolpidem on a nightly basis for one year.

DETAILED DESCRIPTION:
The acknowledged drugs of choice for the pharmacological treatment of insomnia are the benzodiazepine receptor agonist hypnotics (BzRA). Studies show that at therapeutic doses, used over the short-term, the abuse liability of BzRAs is relatively low and their efficacy outweighs their minimal risks. However, an increasing number of patients use BzRAs nightly for longer periods of time than is currently indicated (i.e. 4 weeks) and, minimal data on the long-term abuse liability and efficacy of these drugs exist.

This project, using both prospective and retrospective methods, will address questions about the long-term abuse liability and efficacy of the BzRAs. The questions being raised are: What are the abuse liability and efficacy of hypnotics currently being used chronically and what is the prospective abuse liability and efficacy of hypnotics used chronically? Zolpidem is the chosen standard for this project as it is the most frequently prescribed BzRA and also arguably the BzRA with the best short-term efficacy and safety profile. The focus of the first question is clinical; it is about the long-term abuse liability and efficacy of BzRAs, specifically zolpidem, as it is currently being prescribed and about the type of patients who receive this drug. The second question addresses the issue of whether a standard BzRA can be prescribed efficaciously and safely for the long-term to patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-70 yrs
2. non-pregnant females who agree to standard birth control for 12 months and males
3. two of the following chronic insomnia complaints: >30 min sleep latency, < 6 hrs sleep, or nonrestorative sleep.
4. meet DSM-IV criteria for primary insomnia

Exclusion Criteria:

1. any acute or unstable illness: conditions making it unsafe for the subject to participate, conditions with a potential to disturb sleep (i.e. acute pain, respiratory infection), and conditions which could interact with the pharmacokinetics or pharmacodynamics of zolpidem.
2. chronic illnesses: renal failure, liver disease, seizures, and dementing illnesses.
3. current psychiatric diseases: alcohol or substance abuse, depression, and schizophrenia.
4. a history of alcohol or substance abuse within the past two years.
5. a prestudy positive urine drug screen
6. consuming >14 standard (1oz) alcoholic drinks per week
7. caffeine consumption >300 mg/day
8. smoking during the night (11pm-7am).
9. medications including: anxiolytics, hypnotics. both prescription and OTC, (except in the chronic zolpidem group), antidepressants, anticonvulsants, sedating H1 antihistamines (non-sedating second generation H1 antihistamines are allowed), systemic steroids, respiratory stimulants and decongestants, prescription and OTC stimulants, prescription and OTC diet aids, herbal preparations, and narcotic analgesics. All medications and doses will be documented.
10. sleep disordered breathing (SDB) defined as >10 apnea-hypopneas events per hour of sleep time or any other primary sleep (e.g., restless legs syndrome) or circadian disorder.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary insomniacs meeting DSM-IV criteria, ages 23-70 yrs. old, were recruited from public advisement for a double-blind placebo controlled study. Participants were in good general health as determined by a physical exam and laboratory tests. The Structured Clinical Interview for DSM Disorders (SCID) and the Hamilton Depression Scale were used to exclude those with psychiatric disorders, drug, and alcohol dependence. To confirm the absence of illicit drugs, participants underwent a urine drug screen. Additionally, participants had a screening sleep efficiency of <85% on an 8-hr nocturnal polysomnogram (NPSG) and had no primary sleep disorders. Pregnant or lactating females were excluded from study participation.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2005-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sleep recording measures | one year

SECONDARY OUTCOMES:
Urine and saliva cortical levels | one year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A. Roehrs, Ph.D., Principal Investigator — Henry Ford Health System; Surilla Randall, Ph.D., Study Director — Henry Ford Health System
Locations (1):
- Henry Ford Sleep and Research Center, Detroit, Michigan, United States

REFERENCES:
- [Result] Roehrs TA, Randall S, Harris E, Maan R, Roth T. Twelve months of nightly zolpidem does not lead to rebound insomnia or withdrawal symptoms: a prospective placebo-controlled study. J Psychopharmacol. 2012 Aug;26(8):1088-95. doi: 10.1177/0269881111424455. Epub 2011 Oct 16. PMID 22004689
- [Result] Roehrs TA, Randall S, Harris E, Maan R, Roth T. Twelve months of nightly zolpidem does not lead to dose escalation: a prospective placebo-controlled study. Sleep. 2011 Feb 1;34(2):207-12. doi: 10.1093/sleep/34.2.207. PMID 21286241
- [Derived] Roehrs T, Roth T. Hyperarousal in insomnia: pre-sleep and diurnal cortisol levels in response to chronic zolpidem treatment. Sleep Med. 2019 Sep;61:52-56. doi: 10.1016/j.sleep.2019.04.010. Epub 2019 Apr 25. PMID 31255482
- [Derived] Roehrs TA, Roth T. Hyperarousal in insomnia and hypnotic dose escalation. Sleep Med. 2016 Jul;23:16-20. doi: 10.1016/j.sleep.2016.06.008. Epub 2016 Jul 6. PMID 27692272
- [Derived] Roehrs TA, Roth T. Gender Differences in the Efficacy and Safety of Chronic Nightly Zolpidem. J Clin Sleep Med. 2016 Mar;12(3):319-25. doi: 10.5664/jcsm.5574. PMID 26446253
- [Derived] Randall S, Roehrs TA, Roth T. Efficacy of eight months of nightly zolpidem: a prospective placebo-controlled study. Sleep. 2012 Nov 1;35(11):1551-7. doi: 10.5665/sleep.2208. PMID 23115404